CLINICAL TRIAL: NCT01255527
Title: A Phase 1/2, Open-label, Prospective, Multicenter Study to Evaluate the Efficacy and Safety of the Lower Dose of Bortezomib Plus Busulfan and Melphalan as a Conditioning Regimen in Patients With Multiple Myeloma Undergoing Autologous Peripheral Blood Stem Cell Transplantation- KMM103 Study
Brief Title: Evaluating the Efficacy and Safety of the Lower Dose of Bortezomib Plus Busulfan and Melphalan as a Conditioning Regimen in Patients With Multiple Myeloma Undergoing Autologous Peripheral Blood Stem Cell Transplantation- KMM103 Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2010-0482
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Multiple Myeloma Patients Who Candidate for Autologous Peripheral Blood Stem Cell Transplantation
MeSH Terms: interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Busulfan (Active Comparator)
  Interventions: Drug: Bortezomib
- Melphalan (Active Comparator)
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Bortezomib i.v. 0.7, 1.0 and 1.3 mg/m²/day
  Other Names: VELCADE®

SUMMARY:
Despite the advantages of autologous stem cell transplantation (ASCT) over conventional chemotherapy,1,2 the results of high-dose chemoradiotherapy in multiple myeloma (MM) are still unsatisfactory with a 6-year event free survival (EFS) of only 24%.

Based on existing data, bortezomib-containing regimens are currently accepted at many centers as an induction treatment option for patients with symptomatic MM, particularly if it is planned to offer subsequent high-dose therapy with ASCT. So we will use bortezomib-containing regimens as induction prior to this novel conditioning regimen. The objective of the present study is to compare the toxicity and therapeutic efficacy of a new high-dose regimen using dose-escalation of BOR, BU and MEL for ASCT in the Korean patients with MM. The patients should be treated with bortezomib-containing regimens as an induction therapy before ASCT. We will specifically analyze (i) the efficacy of the conditioning regimen in improving the pre-ASCT status, response rate (ii) engraftment and transplant-related mortality (TRM) and (iii) the impact on survival including progression-free survival (PFS) and overall survival (OS).

Triple combination of conditioning will enhance the response rate after ASCT, and will improve not only PFS, but also OS. We think that data from this study may further strengthen feasibility of BOR in conditioning prior to ASCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of multiple myeloma (MM)
* Symptomatic MM (multiple myeloma with related organ or tissue damage)
* The MM patients with induction chemotherapy with bortezomib-containing regimens (bortezomib±steroid±adrimycin)
* The MM patients who performed the peripheral blood stem cell collection and appropriate stem cell counts (CD34+ cells 2 x 106/kg).
* Age 20-65 years
* Performance status: ECOG (Eastern Cooperative Oncology Group) 0-2.
* Patient has measurable disease, defined as follows: measurable disease is defined as serum M-protein ≥ 1 g/dL or urine M-protein ≥ 200 mg/24 hours when the patients started the primary induction therapy.
* Cardiac ejection fraction ≥ 50 % as measured by MUGA or 2D ECHO without clinically significant abnormalities
* Adequate liver functions: - Transaminase (AST/ALT) < 3 X upper normal value - Bilirubin < 2 X upper normal value
* Adequate hematological function: Platelet count ≥ 75 x 109/L, hemoglobin ≥ 8 g/dL, (Prior RBC transfusion or recombinant human erythropoietin use is allowed), absolute neutrophil count (ANC) ≥ 1.0 x 109/L
* A negative serum or urine pregnancy test prior to treatment must be available both for pre menopausal women and for women who are < 1 years after the onset of menopause.
* Expected survival 6 months
* Informed consent

Exclusion Criteria:

* Systemic AL amyloidosis, smoldering multiple myeloma or MGUS.
* Patient with plasma cell leukemia (> 20% plasma cells in the PB and an absolute plasma cell count of at least 2000/μL)
* Patients who received an extensive radiation therapy within 4 weeks
* Patient is known to be Human Immunodeficiency Virus (HIV) positive.
* Patient has known clinically active Hepatitis B or C.
* Previous renal transplantation
* Severe peripheral neuropathy (Grade 2 or higher as defined by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 3.0)
* Any other malignancies within the past 5 years except curatively treated non-melanoma skin cancer or in situ carcinoma of cervix uteri
* Pregnant or lactating women, women of childbearing potential not employing adequate contraception
* Other serious illness or medical conditions i. Uncontrolled or severe cardiovascular disease, including myocardial infarction, within 6 months of enrollment, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, clinically significant pericardial disease, or cardiac amyloidosis ii. History of significant neurological or psychiatric disorders including dementia or seizures iii. Active uncontrolled infection (viral, bacterial or fungal infection) iv. Active ulcers detected at gastroscopy v. Other serious medical illnesses
* Known hypersensitivity to any of the study drugs or its ingredients (i.e., hypersensitivity to compounds containing boron or mannitol)
* Concomitant administration of any other experimental drug under investigation, or concomitant chemotherapy, hormonal therapy, or immunotherapy.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2010-10; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Maximally tolerated dose (Phase 1) | 28 days

SECONDARY OUTCOMES:
CR and near CR (Phase 2) | 3 months

CONTACTS AND LOCATIONS:
Locations (8):
- South Korea (8):
  - National Cancer Center, Goyang
  - Gachon University Gill Hospital, Incheon
  - Severance Hospital, Seoul
  - ASAN Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul